CLINICAL TRIAL: NCT03095820
Title: A 12-week Multidomain Intervention With Contingency Management for Older Adults With Major Depressive Disorder: A Community-based Randomized Clinical Trial
Brief Title: Multidomain Intervention for Older Adults With Major Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Sang Joon Son, Assistant Professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AJIRB-SBR-SUR-15-132
Record Dates: First submitted 2017-03-21; First posted 2017-03-30 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Major Depressive Disorder
Keywords: Community; Depressive Symptoms; Mental Health Program; Older adults
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: Randomized controlled parallel-design study
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention, we were unable to blind the nurses performing the intervention. However, to achieve double blinding as rigorously as possible, group allocation was not divulged to participants, and symptoms were rated by independent psychologists unaware of the randomization status.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supportive therapy (Active Comparator): The control group received supportive therapy for 12 weeks. In addition to a telephone call once a week and a home visit once a month, this program consisted of identification of physical problems, encouragement of general exercise, encouragement of pleasant activities, and so forth. The control program did not feature any specific goal setting by the participants, specific education about the benefits of achievement of such goals, or symbolic prizes.
  Interventions: Behavioral: Supportive therapy
- Multidomain intervention (Experimental): As a multidomain intervention, four evidence-based therapeutic approaches (physical activity, healthy diet, social activity, and emotional regulation) were incorporated into the program.
  In terms of the healthy diet intervention, we encouraged participants to perform at least 30 min of above-moderate physical activity, three times per week. In terms of the healthy diet intervention, the intervention consisted of encouraging participants to consume high quantities of fish, olive oil, legumes, vegetables, and fruit, at a frequency of at least twice a week. In terms of the social activity intervention, we encouraged participants to participate in social organizations, such as the senior center, the hall of the elderly, a fraternity, a reunion, and a clan gathering, at least once a week. In terms of the emotional regulation intervention, we a performed brief cognitive restructuring task for 20 min per visit.
  Interventions: Behavioral: Multidomain intervention

INTERVENTIONS:
Behavioral: Supportive therapy
  Arms: Supportive therapy
Behavioral: Multidomain intervention
  Arms: Multidomain intervention

SUMMARY:
To assess the effectiveness of a 12-week multidomain intervention with contingency management for reducing depressive symptoms in older adults with major depressive disorder.

DETAILED DESCRIPTION:
Awareness of the necessity and importance of community-based multidomain psychosocial intervention for late-life depression has increased. However, few studies have attempted to integrate several therapeutic approaches in one intervention program.

Main objective of this study is to assess the effectiveness of a 12-week multidomain intervention with contingency management for reducing depressive symptoms in older adults with major depressive disorder.

We plan to conduct a randomized controlled parallel-design study. We plan to allocate study participants to multidomain intervention or supportive therapy group, in a 1:1 ratio. Block randomization using SAS (PLAN procedure) and sample size estimation were performed. We estimated that, with at least 40 participants per group and an attrition rate of 10%, we could achieve a power of at least 0.80 (beta = 0.2, two-tailed alpha = 0.05).

Intervention was based on the financial and human resources of a community mental health service, and involved four home visits and 12 telephone calls over 12 weeks. Four evidence-based therapeutic approaches (physical activity, healthy diet, social activity, and emotional regulation) were incorporated into the multidomain intervention program. To maintain participant motivation, we plan to apply contingency management based on operant conditioning theory.

The primary outcome is the change in depressive symptoms, as measured by the Montgomery-Asberg Depression Rating Scale (MADRS). Secondarily, we plan to investigate changes in resting-state functional connectivity in the default mode, salience, and central executive networks.

ELIGIBILITY:
Inclusion Criteria:

1. a diagnosis of non-psychotic, unipolar major depressive disorder, based on the Mini-International Neuropsychiatric Interview
2. a Montgomery-Asberg Depression Rating Scale (MADRS) score of 17 or higher
3. the use of antidepressants at stable dosage for at least 6 weeks prior to study entry, without any recommendation for changes in medication for the 12 weeks of the intervention. Pharmacotherapy was uncontrolled and was provided by physicians.

Exclusion Criteria:

1. a history of psychiatric disorder (mental retardation, schizophrenia, bipolar disorder, and dementia)
2. a history of neurological disorder, such as brain tumor, intracranial hemorrhage, subarachnoid hemorrhage, epilepsy, hydrocephalus, encephalitis, metabolic encephalopathy, or other neurologic conditions that could interfere with the study
3. a history of significant hearing or visual impairment
4. a history of physical illnesses that could interfere with the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale(MADRS) | Baseline, 4 weeks, 8 weeks, 12 weeks
  Change from baseline depressive symptoms at 4, 8, 12 weeks

SECONDARY OUTCOMES:
resting-state fMRI | Baseline, 12 weeks
  brain functional connectivity

CONTACTS AND LOCATIONS:
Overall Officials: Sang Joon Son, MD,PhD, Principal Investigator — Ajou Univeristy School of Medicine
Locations (1):
- Ajou University Hospital, Suwon, Gyunggi-do, South Korea

REFERENCES:
- [Derived] Roh HW, Hong CH, Lim HK, Chang KJ, Kim H, Kim NR, Choi JW, Lee KS, Cho SM, Park B, Son SJ. A 12-week multidomain intervention for late-life depression: a community-based randomized controlled trial. J Affect Disord. 2020 Feb 15;263:437-444. doi: 10.1016/j.jad.2019.12.013. Epub 2019 Dec 9. PMID 31969275